CLINICAL TRIAL: NCT02332928
Title: Melatonin Supplementation for Cancer-related Fatigue in Patients Receiving Radiotherapy: A Double Blind Placebo-Controlled Trial
Brief Title: Melatonin Supplementation for Cancer-related Fatigue in Patients Receiving Radiotherapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MCC-12-08248; HM20003275 (Other: IRB); NCI-2015-00345 (Registry Identifier: CTRP); P30CA016059 (NIH)
Record Dates: First submitted 2014-12-16; First posted 2015-01-07 (Estimated); Results first posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer - Female
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 20 mg Melatonin (Active Comparator): RT (as clinically indicated) + melatonin (Subjects will receive 20-mg oral melatonin the night before their first RT treatment, each night throughout the course of RT treatment, and for 2 weeks following the completion of RT).
  Interventions: Drug: Melatonin
- Placebo (Placebo Comparator): RT (as clinically indicated) + placebo (Subjects will receive 20-mg oral placebo the night before their first RT treatment, each night throughout the course of RT treatment, and for 2 weeks following the completion of RT).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Melatonin — Melatonin + RT (as clinically indicated) (Subjects will receive 20-mg oral melatonin or placebo the night before their first RT treatment, each night throughout the course of RT treatment, and for 2 weeks following the completion of RT).
  Arms: 20 mg Melatonin
Drug: Placebo — Placebo + RT (as clinically indicated) (Subjects will receive 20-mg oral melatonin or placebo the night before their first RT treatment, each night throughout the course of RT treatment, and for 2 weeks following the completion of RT).
  Arms: Placebo

SUMMARY:
This is a double-blind, placebo-controlled trial wherein subjects with breast cancer will be randomized to receive either 20 mg oral melatonin or placebo the night before their first radiotherapy (RT), nightly throughout their RT, and for an additional 2 weeks following the completion of their RT. After informed consent is obtained from eligible subjects, they will then be electronically randomized on a 1:1 ratio to melatonin treatment or placebo. The subjects will be stratified according to treatment duration (less than 3 weeks; equal to or greater than 3 weeks) and prior chemotherapy.

DETAILED DESCRIPTION:
Subjects will be randomized to receive either melatonin or placebo. Subjects will receive 20-mg oral melatonin or placebo the night before their first RT treatment, each night throughout the course of RT treatment, and for 2 weeks following the completion of RT. Patients with localized breast cancer will receive standard-of-care RT as determined by the treating physician. The RT regimens include: (1) 1 week of accelerated (APBI); (2) 3-4 weeks of an accelerated hypofractionation RT schedule; and (3) 6-8 weeks of a standard RT schedule. No additional concomitant medication or supportive care guidelines are required for this study. Subjects will receive daily melatonin or placebo beginning the night before their course of RT and for an additional 2-week period that extends beyond the conclusion of their RT. Subjects will be given a Study Diary to record their use of study medication. Patients will be followed for 60 days after removal from the study treatment or until death, whichever occurs first. Patients removed from the study treatment for unacceptable adverse events (AEs) will be followed until resolution or stabilization of the adverse event.

ELIGIBILITY:
Inclusion Criteria

1. Ambulatory outpatients with breast (including ductal carcinoma in situ [DCIS]) cancer.
2. Patients to be treated with RT for curative intent.
3. Women ≥18 years of age.
4. Eastern Cooperative Oncology Group (ECOG) performance status <3 (Appendix 4).
5. Hemoglobin ≥ 9 g/dL
6. Either post-menopausal, surgically sterilized, or willing to use an acceptable method of birth control during study treatment and for 3 months afterwards.
7. Subjects who are currently taking melatonin must discontinue melatonin for 5 days before enrolling in the study.
8. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria

1. Fatigue brought on by conditions other than cancer such as (the indicated tests are required only if that mechanism of fatigue is suspected):

   * uncontrolled hypothyroidism (TSH >10 IU)
   * hypercalcemia (calcium >11 mg/dL) Calcium (Ca) = Serum Calcium (SerumCa) + 0.8 * (NormalAlbumin - PatientAlbumin)
   * decompensated congestive heart failure
   * chronic obstructive pulmonary disease requiring oxygen replacement
2. Patients with a creatinine clearance <30 mL/min
3. Aspartate aminotransferase (AST) > 3X upper limit of normal (ULN)
4. Alanine aminotransferase (ALT) > 3X ULN
5. Bilirubin > 1X ULN
6. Use of systemic steroids, or other pharmacological agents such as methylphenidate for cancer-related fatigue
7. Current use of American ginseng, remelteon, or warfarin.
8. Depression ≥ grade 2 (CTCAE v4.0)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-03-25 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo I Urdaneta, MD, Principal Investigator — Massey Cancer Center
Locations (1):
- Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 20 mg Melatonin | Placebo
Started | 40 | 40
Completed | 39 | 38
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Cronavirus disease (COVID-19) Precautions | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 20 mg Melatonin | Placebo | Total
Number analyzed (Participants) | 39 | 38 | 77
Age, Customized [Median (Full Range); unit: years] | 54 [35 to 73] | 58 [38 to 78] | 56.5 [35 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 38 | 77
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 39 | 37 | 76
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 11 | 21
  White | 27 | 27 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 39 | 38 | 77

OUTCOME MEASURES:

1. Primary Outcome: Comparison of FACIT-Fatigue Subscale
Description: Determine if the average increase in fatigue (as measured by the Functional Assessment of Chronic Illness Therapy (FACIT-Fatigue subscale) from baseline to completion of RT is different in those patients who received melatonin than in those who received placebo. The FACIT-F is a well-validated QOL instrument widely used for the assessment of cancer-related fatigue in clinical trials. It consists of 27 general QOL questions divided into 4 domains (physical, social, emotional, and functional), plus a 13-item fatigue sub-score. The patient rates the intensity of fatigue and its related symptoms on a scale of 0-4. The total score ranges between 0 and 52, with higher scores denoting less fatigue.
Time Frame: Baseline,( Day 1), 2 weeks post radiation therapy completion (variable, approximately 58 weeks)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | 20 mg Melatonin | Placebo
Number analyzed (Participants) | 39 | 38
score on a scale | -4.39 (1.24) | 0.74 (1.69)

2. Secondary Outcome: Comparison of Functional Assessment of Chronic Illness Therapy (FACIT-F) Scores in Fatigue From Baseline Until 2 Weeks After Completion of RT in Those Patients Who Received Melatonin Compared to Those Who Received Placebo.
Description: Determine whether the average increase in fatigue from baseline until 2 weeks after completion of RT is less in those patients who received melatonin than in those who received placebo. The FACIT-F is a well-validated QOL instrument widely used for the assessment of cancer-related fatigue in clinical trials. It consists of 27 general QOL questions divided into 4 domains (physical, social, emotional, and functional), plus a 13-item fatigue sub-score. The patient rates the intensity of fatigue and its related symptoms on a scale of 0-4. The total score ranges between 0 and 52, with higher scores denoting less fatigue.
Time Frame: Baseline,( Day 1), 2 weeks post radiation therapy completion (variable, approximately 58 weeks)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | 20 mg Melatonin | Placebo
Number analyzed (Participants) | 39 | 38
score on a scale | -2.78 (1.5) | 1.3 (1.97)

3. Secondary Outcome: Comparison in Functional Assessment of Chronic Illness Therapy (FACIT) in Fatigue From Baseline Until 8 Weeks After Completion of RT in Those Patients Who Received Melatonin Compared to Those Who Received Placebo.
Description: Determine whether the average increase in fatigue from baseline until 8 weeks after completion of RT is less in those patients who received melatonin than in those who received placebo. The FACIT-F is a well-validated QOL instrument widely used for the assessment of cancer-related fatigue in clinical trials. It consists of 27 general QOL questions divided into 4 domains (physical, social, emotional, and functional), plus a 13-item fatigue sub-score. The patient rates the intensity of fatigue and its related symptoms on a scale of 0-4. The total score ranges between 0 and 52, with higher scores denoting less fatigue.
Time Frame: Baseline (Day 1) and 8 weeks post RT (variable, approximately 64 weeks)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | 20 mg Melatonin | Placebo
Number analyzed (Participants) | 39 | 38
score on a scale | 0.65 (1.31) | 4.58 (1.26)

4. Secondary Outcome: Comparison of Edmonton Symptom Assessment System (ESAS) Scores Obtained at Baseline Until Completion of RT.
Description: Average increase in symptoms from baseline until completion of RT for those patients who received melatonin compared to those who received placebo. The ESAS assesses 10 symptoms experienced by cancer patients during the previous 24 hours: pain, fatigue, nausea, depression, anxiety, drowsiness, dyspnea, anorexia, sleep disturbance, and feelings of well-being. The severity of each symptom is rated on a numerical scale of 0-10 (0 = no symptom, 10 = worst possible severity).
Time Frame: Baseline,( Day 1), 2 weeks post radiation therapy completion (variable, approximately 58 weeks)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | 20 mg Melatonin | Placebo
Number analyzed (Participants) | 39 | 38
score on a scale
  Change in Anxiety | -0.26 (0.48) | -0.69 (0.32)
  Change in Best Well Being | 0.29 (0.3) | 0.41 (0.49)
  Change in Depression | -2 (0.21) | -0.34 (0.31)
  Change in Drowsiness | 1.39 (0.39) | 0.81 (0.48)
  Change in Lack of Appetite | 0.35 (0.49) | 0.47 (0.29)
  Change in Nausea | 0.19 (0.14) | 0.06 (0.15)
  Change in Pain Score | 0.74 (0.45) | 1.48 (0.52)
  Change in Shortness of Breath | -0.29 (0.26) | -0.44 (0.18)
  Change in Sleep | 0.93 (0.38) | -0.07 (0.62)
  Change in Tiredness | 1.81 (0.41) | 0.28 (0.51)

5. Secondary Outcome: Comparison of the Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue-Short Form 8a Scores Obtained at Baseline and at the Completion of RT.
Description: Determine whether the average increase in fatigue (as measured by the PROMIS Fatigue-Short Form 8a) from baseline to completion of RT is less in those patients who received melatonin compared to those who received placebo. The higher score, the worse fatigue. The PROMIS Fatigue-Short Form 8a scale consists of 8 general questions regarding fatigue. The patient rates the intensity of fatigue and related symptoms on a scale of 1-5. The total score can range between 8 and 40, with higher scores denoting more fatigue.
Time Frame: Baseline,( Day 1), 2 weeks post radiation therapy completion (variable, approximately 58 weeks)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | 20 mg Melatonin | Placebo
Number analyzed (Participants) | 39 | 38
score on a scale | 3.51 (1.08) | -0.52 (1.2)

6. Secondary Outcome: Determine the Level of Agreement in Reported Fatigue Scores When 2 Different Survey Instruments Are Used to Measure Fatigue.
Description: Compare the scores obtained with the FACIT-Fatigue subscale and the PROMIS Fatigue-Short Form at completion of RT. The FACIT-F is a well-validated QOL instrument widely used for the assessment of cancer-related fatigue in clinical trials. It consists of 27 general QOL questions divided into 4 domains (physical, social, emotional, and functional), plus a 13-item fatigue sub-score. The patient rates the intensity of fatigue and its related symptoms on a scale of 0-4. The total score ranges between 0 and 52, with higher scores denoting less fatigue. The PROMIS Fatigue-Short Form 8a scale. It consists of 8 general questions regarding fatigue. The patient rates the intensity of fatigue and related symptoms on a scale of 1-5. The total score can range between 8 and 40, with higher scores denoting more fatigue.
Time Frame: Baseline,( Day 1), 2 weeks post radiation therapy completion (variable, approximately 58 weeks)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | 20 mg Melatonin | Placebo
Number analyzed (Participants) | 40 | 38
score on a scale
  FACIT | -4.39 (1.24) | 0.74 (1.69)
  PROMIS | 3.51 (1.08) | -0.52 (1.2)

7. Secondary Outcome: Compare the Number of Hospital Admissions, Emergency Center Visits, and Medical Days Off Work Between Patients Receiving Melatonin Compared to Placebo.
Description: Determine whether patients receiving melatonin have fewer hospital admissions, emergency center visits, and medical days off work than patients receiving placebo
Time Frame: Baseline (day 1) to 8 weeks post RT (variable, approximately 64 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | 20 mg Melatonin | Placebo
Number analyzed (Participants) | 39 | 38
Participants
  Emergency Department Visit | 6 | 3
  Hospital Admission | 7 | 5
  Medical Day Off From Work | 15 | 4

ADVERSE EVENTS:
Time Frame: 30 days following completion of treatment, an average of 20 weeks.
Arm/Group | 20 mg Melatonin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/39 | 1/38
Serious Adverse Events (participants affected / at risk) | 0/39 | 3/38
Other Adverse Events (participants affected / at risk) | 37/39 | 37/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20 mg Melatonin (N=39) | Placebo (N=38)
Creatinine Increased (Investigations) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Nervous System Disorders-Other, specify (Nervous system disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20 mg Melatonin (N=39) | Placebo (N=38)
Anemia (Blood and lymphatic system disorders) | 37 (440) | 37 (346)
Restrictive Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 12 (16) | 8 (10)
Constipation (Gastrointestinal disorders) | 4 (4) | 1 (1)
Dental Caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (4) | 3 (5)
Dysphagia (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 2 (3) | 1 (1)
Gastrointestinal Disorders- Other, specified (Gastrointestinal disorders) | 2 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 10 (13) | 12 (15)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (3)
Edema Face (General disorders) | 1 (1) | 0 (0)
Edema Limbs (General disorders) | 2 (4) | 0 (0)
Fatigue (General disorders) | 32 (64) | 31 (53)
Flu Like Symptoms (General disorders) | 1 (1) | 0 (0)
General Disorders and Administration Site Conditions-Other Specified (General disorders) | 5 (5) | 1 (1)
Localized Edema (General disorders) | 1 (1) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 1 (2) | 0 (0)
Pain (General disorders) | 10 (15) | 8 (12)
Breast Infection (Infections and infestations) | 1 (3) | 0 (0)
Dermatitis Radiation (Injury, poisoning and procedural complications) | 25 (41) | 27 (40)
Alkaline Phosphatase Increased (Investigations) | 0 (0) | 1 (1)
Creatinine Increased (Infections and infestations) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Joint Range of Motion Decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Musculoskeletal and connective Tissue Disorder - Other, Specify (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (39) | 2 (3)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Dizziness (Nervous system disorders) | 16 (22) | 9 (14)
Dysgeusia (Nervous system disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 21 (35) | 15 (26)
Nervous System Disorder-Other, Specify (Nervous system disorders) | 2 (2) | 2 (2)
Peripheral Sensory Neuropathy (Nervous system disorders) | 4 (4) | 1 (1)
Somnolence (Nervous system disorders) | 27 (45) | 21 (34)
Anxiety (Psychiatric disorders) | 18 (29) | 15 (19)
Confusion (Psychiatric disorders) | 7 (12) | 5 (6)
Depression (Psychiatric disorders) | 16 (24) | 18 (29)
Insomnia (Psychiatric disorders) | 6 (9) | 4 (7)
Irritability (Psychiatric disorders) | 9 (9) | 1 (1)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 2 (2) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Breast Pain (Reproductive system and breast disorders) | 7 (9) | 7 (8)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pain of Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (5)
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 5 (5) | 7 (8)
Skin Hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Ulceration (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Hot Flashes (Vascular disorders) | 4 (4) | 4 (5)
Hypertension (Vascular disorders) | 3 (4) | 3 (3)
Lymphedema (Vascular disorders) | 1 (1) | 3 (5)

LIMITATIONS AND CAVEATS:
The study had an initial goal of 142 patients, with interim analysis at half recruitment. Upon recommendation from the Data and Safety Monitoring Committee (DSMC), the study concluded at interim analysis due to lack of efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-10): https://cdn.clinicaltrials.gov/large-docs/28/NCT02332928/Prot_SAP_001.pdf
  • Informed Consent Form (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/28/NCT02332928/ICF_000.pdf